CLINICAL TRIAL: NCT04009239
Title: Time Restricted Feeding and Metabolic Rhythms
Acronym: Rhythm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16-2754; K01DK113063 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Diabetes
Keywords: Weight loss; Diet
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Time Restricted Feeding (Experimental): Consume meals for 7 days during an 8 hour window starting 1 hour after habitual wake time.
  Interventions: Behavioral: Time Restricted Feeding
- Mid-day Time Restricted Feeding (Experimental): Consume meals for 7 days during an 8 hour window starting 6 hours after habitual wake time.
  Interventions: Behavioral: Time Restricted Feeding

INTERVENTIONS:
Behavioral: Time Restricted Feeding — Consuming energy during a short interval during the day

SUMMARY:
Current guidelines for the prevention and treatment of obesity focus on caloric restriction diets and increasing physical activity, but long-term compliance to these strategies is poor. The timing of meal intake relative to the light-dark and sleep-wake cycle is rarely considered in metabolic health; and modifying meal timing is likely easier to implement in daily life than reducing caloric intake and/or increasing physical activity. This project will test whether restricting the timing of energy intake to a short-defined period during wakefulness can be used to improve fuel utilization patterns and enhance circadian rhythms in metabolic tissues to optimize health.

DETAILED DESCRIPTION:
Time restricted feeding (TRF; eating within <10-h period followed by >14-h fast) is a promising meal timing paradigm that in rodent studies improves multiple health indicators. When provided access to a high-fat diet ad libitum, mice rapidly gain weight. However, when fed the same diet under TRF conditions (food access restricted to an 8-h window during the active phase) mice appear to be protected from excessive weight gain and metabolic diseases. Preliminary studies in humans are showing improvements in 24-h glucose variability, fat oxidation, and blood pressure with TRF aligned to the early portion of the day compared to the ad libitum feeding schedule. A major research gap is whether the timing of the feeding window relative to sleep modifies metabolic responses. In a recent pilot and feasibility study incorporating TRF into a weight loss intervention the researchers asked participants to consume all food within a 10-h window to starting 1-h after waking for 12-weeks. The researchers' design choice was based on data showing that consuming energy in the evening is related to a two-fold increase in obesity risk. There also appears to be reduced weight loss effectiveness in dieters who consume the main meal later in the day. Some of the participants in the weight loss trial reported difficulty adhering to the early feeding schedule because it does not align well with social schedule (e.g., eating dinner with the family in the evening). Therefore, an important clinical question is whether late or mid-day TRF will result in similar metabolic benefits compared to the early TRF paradigm that has been tested in other studies.

Additional rationale for studying early vs. late timed feeding is to address a fundamental question, "can timed meals shift the timing of metabolic rhythms?". Peripheral circadian clocks located in liver, adipose, and muscle tissue are sensitive to meal timing and control daily oscillations in fuel utilization and storage. A small study of 8 men demonstrated that a 5-h delay and meal timing was sufficient to delay the rhythmic expression of clock genes in white adipose tissue. Therefore, the investigators will leverage the design of the present study to examine the impact of meal timing on peripheral circadian rhythms in metabolism and their alignment to the sleep cycle.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with overweight and class I obesity (N=12, Age=20-50 years; BMI 25-35 kg/m2)
* Low physical activity level (≤150 min/wk of moderate-to-vigorous activity);
* For Females- Not currently pregnant or lactating and not pregnant within the past 6 months
* Habitually consume food over a window of >12 h/day;
* Pass a medical and physical screening performed by the study physician.
* Report a habitual, regular sleep-wake cycle for the month preceding screening that involved going to bed between 2200 and 0100h and getting up between 0600 and 0900 h with >7 h and <9.25 h in bed;
* Agree to eat control diets at imposed times for 1 week prior to the inpatient CTRC visits;
* Agree to keep a regular sleep/wake schedule for the duration of the study
* Possess a smart phone to install and utilize the meal timing application.

Exclusion Criteria:

* Subjects must not be currently participating in another research study that would influence their safe participation in this study. For example, subjects must not be participating in a research study in which they ingest experimental medication, or which involves blood samples, since both of these factors could increase risk of participation;
* Being considered unsafe to participate as determined by the study physician;
* Taking medications affecting weight, triglycerides, energy intake/energy expenditure, or sleep in the last 3 months;
* Having abnormal blood chemistry and/or hematology as deemed significant by the study physician;

  o Have one or more of the following out-of-range values measured on a fasting blood sample: glucose > 126 mg/dl, HbA1c > 6.5%, thyroid stimulating hormone <0.5 or >5.0 uU/ml. Subjects who may be anemic (hemoglobin <14.5 g/dl men, <12.3 g/dl women), have abnormal liver function tests (alanine amino transferase > 47 U/l, aspartate aminotransferase, > 47 U/l, alkaline phosphatase <39 or >117 U/l) or creatinine (>1.1 mg/dl)
* Significant abnormality in clinical laboratory values
* Ever having a history of systemic, psychiatric, neurological disease, or drug and alcohol abuse;
* History of cardiovascular disease, diabetes, uncontrolled hypertension, untreated thyroid, renal, hepatic diseases, dyslipidemia or any other medical condition affecting weight or lipid metabolism;
* Score > 18 on Beck Depression Index (BDI) will require further assessment by the study physician to determine if it is appropriate for the subject to participate in the study;
* Use of a continuous positive airway pressure (CPAP) device for the treatment of obstructive sleep apnea (OSA). A score of >10 on the Epworth sleepiness scale or >5 on the Pittsburgh Sleep Quality Index will require further assessment by the study physician to determine if it is appropriate for the subject to participate in the study;
* Being positive for human immunodeficiency virus or hepatitis B or C;
* Being a smoker or having been a smoker in the previous 6 months;
* Abnormal eating patterns identified by registered dietician interview (dietary fat<15%, dietary fat>45%, dietary protein >30%);
* Working night shifts;
* Night eating syndrome (at least 25% of food intake is consumed after the evening meal and/or at least two episodes of nocturnal eating per week);
* Traveling > 2 time zones 2 weeks prior to an inpatient CTRC study visit;
* Currently participating in any formal weight loss or physical activity programs or clinical trials.
* Having a clinically significant allergy (e.g., to food stuffs such as shellfish, peanuts);
* Celiac disease or known sensitivity to gluten (the metabolic kitchen is not gluten free certified and cannot accommodate this dietary restriction)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
Total fat oxidation in response to eTRF | Week 1 or Week 5
  Total fat oxidation will measured by whole room calorimetry. Early Time Restricted Feeding (eTRF) may occur at Week 1 or Week 5 depending on randomization.
Total fat oxidation in response to mTRF | Week 1 or Week 5
  Total fat oxidation will measured by whole room calorimetry. Mid-day Time Restricted Feeding (mTRF) may occur at Week 1 or Week 5 depending on randomization.
Insulin sensitivity in response to eTRF | Week 1 or Week 5
  Insulin sensitivity measured by three identical mixed meal tolerance tests administered across the day. Early Time Restricted Feeding (eTRF) may occur at Week 1 or Week 5 depending on randomization.
Insulin sensitivity in response to mTRF | Week 1 or Week 5
  Insulin sensitivity measured by three identical mixed meal tolerance tests administered across the day. Mid-day Time Restricted Feeding (mTRF) may occur at Week 1 or Week 5 depending on randomization.
Glucose control in response to eTRF | Week 1 or Week 5
  Glucose control will be measured by a continuous glucose monitor. Mid-day Time Restricted Feeding (mTRF) may occur at Week 1 or Week 5 depending on randomization.
Glucose control in response to mTRF | Week 1 or Week 5
  Glucose control will be measured by a continuous glucose monitor. Early Time Restricted Feeding (eTRF) may occur at Week 1 or Week 5 depending on randomization.

SECONDARY OUTCOMES:
Difference in dietary fat oxidation between experimental conditions | Week 1 and Week 5
  Dietary fat oxidation will be measured using a stable isotope tracer
Difference in 24h energy expenditure between experimental conditions | Week 1 and Week 5
  24h energy expenditure will be measured using whole room calorimetry
Difference in sleep between experimental conditions | Week 1 and Week 5
  Sleep will be measured by polysomnography
Difference in the melatonin rhythm between experimental conditions | Week 1 and Week 5
  The melatonin profile will be measured in plasma during constant routine protocol
Difference in plasma metabolite rhythms between experimental conditions | Week 1 and Week 5
  Plasma metabolite rhythms will be measured using a constant routine protocol
Difference in plasma hormone rhythms between experimental conditions | Week 1 and Week 5
  Plasma hormone rhythms will be measured using a constant routine protocol
Difference in plasma gene expression rhythms between experimental conditions | Week 1 and Week 5
  Plasma gene expression rhythms will be measured using a constant routine protocol
Difference in energy expenditure rhythms between experimental conditions | Week 1 and Week 5
  Energy expenditure rhythms will be measured by indirect calorimetry during a constant routine protocol
Difference in substrate oxidation rhythms between experimental conditions | Week 1 and Week 5
  Substrate oxidation rhythms will be measured by indirect calorimetry during a constant routine protocol

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Rynders, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717

DOCUMENTS (1):
  • Informed Consent Form (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT04009239/ICF_000.pdf